CLINICAL TRIAL: NCT06287853
Title: A Multi-Center, Prospective Post Market Clinical Follow-Up Evaluating Arthroscopic Rotator Cuff Repair Augmented With TAPESTRY® Biointegrative Implant
Brief Title: Tapestry Rotator Cuff Repair PMCF
Status: Suspended | Type: Observational
Why Stopped: Sponsor has elected to place the Tapestry RC PMCF study on hold. The Tapestry RC product line is being enhanced, and we have chosen to delay data collection on this product until the new devices are available. Study is anticipated to resume in 2026.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: EMBODY-004
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Rotator Cuff Tears; Rotator Cuff Injuries
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Partial Thickness Tear: Patient with a diagnosis of a symptomatic primary partial-thickness tear of the supraspinatus and/or infraspinatus tendons amenable to repair.
  Interventions: Device: Tapestry Biointegrative Implant
- Full Thickness Tear: Patient with a diagnosis of a symptomatic primary full-thickness tear of the supraspinatus and/or infraspinatus tendons amenable to repair.
  Interventions: Device: Tapestry Biointegrative Implant

INTERVENTIONS:
Device: Tapestry Biointegrative Implant — The Tapestry RC Biointegrative Implant System is an arthroscopic delivery and fixation system intended for tendon augmentation with Tapestry Biointegrative Implant during arthroscopic rotator cuff (RC) repair. The system combines the biointegrative collagen-based implant (Tapestry Biointegrative Implant) with bioabsorbable fixation ( Bioabsorbable Anchors). Tapestry Biointegrative Implant is a collagen-based implant composed of type I bovine collagen and poly(D,L-lactide). It is designed to function as a non-constricting, protective layer between the tendon and surrounding tissues.

SUMMARY:
The study design is a prospective, multi-center, single-arm, non-randomized, and noncontrolled post market clinical follow-up study involving orthopedic surgeons skilled in arthroscopic rotator cuff repair as determined by the Sponsor.

DETAILED DESCRIPTION:
The objectives of the study are to calculate the overall clinical success rate, the performance, and clinical benefits, and confirm the safety of the Tapestry RC Biointegrative Implant System.

* The clinical success will be evaluated by absence of rotator cuff re-tear.
* The performance and clinical benefits will be evaluated by functional outcomes measured using standard scoring systems such as the American Shoulder and Elbow Surgeons Shoulder Score (ASES), Visual Analogue Scale (VAS), Constant-Murley Score (CMS), Single Assessment Numeric Evaluation (SANE), Return to Activity, Patient Satisfaction, EQ-5D-5L, and rotator cuff repair outcomes measured using MRI evaluation for repair integrity, quality, tendon tissue thickness and regeneration.
* The safety of the Tapestry RC Biointegrative Implant System will be assessed by monitoring the frequency and incidence of adverse events.

The primary endpoint of this study is defined by the rotator cuff re-tear rate post-operatively. This will be measured against the success criteria of the re-tear rate in 18.3% of cases at two years.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, 21 years and older;
2. Patient with a diagnosis of a symptomatic primary partial-thickness or full-thickness tear of the supraspinatus and/or infraspinatus tendons amenable to repair that meets one of the following criteria:

   * Partial-thickness tear planned for standalone treatment (no surgical repair with sutures/suture anchors) with the Tapestry Biointegrative Implant, or
   * Full-thickness tear planned for treatment with the Tapestry Biointegrative Implant as an adjunct to surgical repair (single or double row repair with sutures/suture anchors);
3. Patient is able and willing to complete the protocol required follow-up;
4. Patient is able and willing to sign the IRB approved informed consent;
5. Independent of study participation, patient qualifies for arthroscopic rotator cuff repair and meets the approved indications for use of the commercially available Tapestry RC Biointegrative Implant System

Exclusion Criteria:

1. Hypersensitivity to bovine-derived materials or poly(D,L-lactide) materials;
2. Patient with an irreparable or partially reparable rotator cuff tear;
3. Revision rotator cuff repair;
4. Off-label use of the study device;
5. Patient is known to be pregnant or nursing;
6. Patient is a prisoner;
7. Patient is a known alcohol or drug abuser;
8. Patient has a psychiatric illness, neurologic disorder, or cognitive deficit that will not allow for proper informed consent or compliance with study requirements;
9. Patient is unable to tolerate magnetic resonance imaging (MRI), due to psychiatric or medical contraindications;
10. Patient is unwilling or unable to give consent or to comply with the follow-up program;
11. Patient has any condition which would in the judgement of the Investigator, place the patient at undue risk or interfere with the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include both males and females undergoing arthroscopic rotator cuff repair due to partial or full-thickness tears of the supraspinatus and/or infraspinatus tendon.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2026-12-28 (Estimated); Primary Completion 2030-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Re-tear rate after arthroscopic rotator cuff repair | 6-month Post-operatively
  Assessed by MRI evaluation at 6 months post-operatively defined using Sugaya classification system.

SECONDARY OUTCOMES:
The American Shoulder and Elbow Surgeons (ASES) Score | Screening/Pre-Op, 6 weeks, 3-month, 6-month, 12-month 24-month Post-operatively
  The American Shoulder and Elbow Surgeon's (ASES) Score is a tool used to measure shoulder function. The ASES score is on a scale of 0 to 100, with 0 being the worst possible score and 100 the best. The score consists of two components - pain and activities of daily living.
Constant-Murley Score (CMS) | Screening/Pre-Op, 6 weeks, 3-month, 6-month, 12-month 24-month Post-operatively
  The Constant-Murley Shoulder Score is a scoring method used by clinicians to assess function of the shoulder. The standard score is on a scale of 0 to 100, with 0 being no shoulder function and 100 being excellent function.
The Single Assessment Numeric Evaluation (SANE) Score | Screening/Pre-Op, 6 weeks, 3-month, 6-month, 12-month 24-month Post-operatively
  The Single Assessment Numeric Evaluation (SANE) Score is a tool used to assess the subject's perception of their affected joint. Participants are requested to rate their shoulder function on a scale of 0 to 100, with 0 as the worst option and 100 being normal shoulder function.
EQ-5D-5L (EuroQol) | Screening/Pre-Op, 6 weeks, 3-month, 6-month, 12-month 24-month Post-operatively
  The 5-level EQ-5D (EQ-5D-5L) is a standardized self-assessed, health related quality of life questionnaire. It is composed of five questions with Likert scale response options (descriptive system) and a visual analog scale (EQ-VAS). The EQ-VAS asks patients to rate their own health from 0 to 100 (the worst and best imaginable health, respectively).
Return to Work/Activity | 6 weeks, 3-month, 6-month, 12-month 24-month post-operatively
  The functional assessment of return to activity is evaluated by the time from discharge to return to work, driving, and sport.
Patient Satisfaction | 6 weeks, 3-month, 6-month, 12-month 24-month Post-operatively
  It is a 5 choice questions asking for patient overall satisfaction to the operative shoulder, from very satisfied to very unsatisfied.
Adverse Event | Screening/Pre-Op, Op, Imme-Post-op, 6 weeks, 3-month, 6-month, 12-month 24-month Post-operatively
  All adverse events reported throughout each subject's length of participation in the study are included.
MRI Sugaya Classification | Screening/Pre-Op, 3-month, 6-month, 12-month 24-month post-operatively
  The Sugaya classification will be used to determine rotator cuff integrity and characterization of retear (symptomatic/asymptomatic, size, shape). Sugaya classifies the integrity of the rotator cuff into five categories: Type I to Type V.
MRI Goutallier Classification | Screening/Pre-Op, 3-month, 6-month, 12-month 24-month post-operatively
  The Goutallier classification will be used to evaluate the rotator cuff quality by classifying the fatty infiltration of the rotator cuff. The Goutallier classification ranges from a grade 0, indicating a completely normal muscles without any fatty streaks, to a grade 4 which indicates more fat is present than muscle

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Premier Ortho & Trauma Specialists, Pomona, California
  - UofL Health, Louisville, Kentucky
  - MedStar Union Memorial Hospital, Baltimore, Maryland